CLINICAL TRIAL: NCT00076700
Title: Enhanced Tactile Memory in the Blind
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040110; 04-N-0110
Record Dates: First submitted 2004-01-31; First posted 2004-02-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Blindness
Keywords: Cross-Modal Plasticity; Functional MRI; Behavior; Memory; Blind; Blindness; Healthy Volunteer; HV
MeSH Terms: conditions — Blindness; Behavior

SUMMARY:
This study will determine if the brain regions in blind people that would normally be involved in vision are used instead to remember touch. Blind people have an enhanced sense of touch compared to sighted people, and they also perform better on tests for certain kinds of memory. This study will examine and compare the results of a touch memory test in blind and sighted people to determine what brain areas are involved in responding to touch.

Blind people and sighted volunteers between 18 and 80 years of age who have no psychiatric problems or neurological problems (other than blindness) may be eligible for this study. Candidates are screened with a medical interview and examination.

Participants undergo one or both of the following procedures:

Behavioral experiment

Sighted participants are blindfolded during this experiment. Subjects sit comfortably in front of a table. They are presented with a number of surfaces placed on a table one at a time and are given 10 seconds to feel each surface with the index finger on their dominant hand. They must concentrate and memorize the surfaces as best they can. After a 15-minute break, they are again presented with a series of surfaces and given 10 seconds to feel each one. This time, they must say as quickly as possibly whether the surface is one they touched previously or is a new surface.

Functional MRI

MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. In this study, subjects undergo MRI scanning of the brain while performing the same touch test described above. For the MRI, the subject lies on a table that slides into the scanner. The MRI machine detects change in the brain regions involved in performing the task.

DETAILED DESCRIPTION:
In the blind, areas of the brain that would normally respond to visual stimuli instead of process information from other sensory modalities such as the somatosensory and auditory domains. Recent studies have shown that the visual cortex of the blind participates in higher-order processing of auditory information including verb generation and retrieval of verbal memories. Because tactile information plays a similarly crucial role when vision is missing (i.e. to read Braille), it has been suggested that the ability to encode and recall tactile information in the blind is superior to that in the sighted.

OBJECTIVES:

The first objective of this protocol is to determine if tactile memory is superior in early blind subjects relative to that in late blind and sighted control subjects.

The second objective is to determine if the visual cortex of blind people can participate in higher-order processing of tactile information such as tactile encoding recognition.

STUDY POPULATION:

Our experiments will make use of early blind, late blind, and sighted control subjects.

DESIGN:

Experiment 1: We will quantify the ability of our study populations to encode into and retrieve from episodic tactile memory. Subjects will be presented with a series of surfaces that they are to palpate and commit to memory, after which they will rest for ten to fifteen minutes. The old surfaces will then be presented again with a same number of new surfaces randomly interleaved. Subjects are to discriminate old from new surfaces.

Experiment 2: We will identify cortical areas associated with successful tactile memory encoding and retrieval in blind individuals and sighted controls using functional magnetic resonance imaging (fMRI). Subjects will perform the memory task from Experiment 1 while in the MRI machine.

OUTCOME MEASURES:

Experiment 1: The primary outcome measure will be recognition memory, a corrected measure of the number of old stimuli correctly remembered.

Experiment 2: The primary outcome measure will be the number of voxels significantly activated in primary visual cortex in early blind subjects as compared to late blind subjects and sighted controls.

We expect the magnitude of visual cortex activation in the early blind during a tactile memory task to correlate with superior performance on the task.

ELIGIBILITY:
INCLUSION CRITERIA:

Early Blind Subjects: Only compliant early blind subjects between the ages of 18 and 80 years who have little to no visual perception due to diseases affecting the peripheral components of the visual system, i.e., blind subjects without any further neurological problems, and with normal MRI brain scans, will be selected.

Late Blind Subjects: Only compliant late blind subjects who have lost their vision after age 4 years due to diseases affecting the peripheral components of the visual system, i.e., blind subjects without any further neurological problems, and with normal MRI brain scans, will be selected.

Sighted controls: Only compliant adult healthy volunteers between the ages of 18 and 80 years with no history of neurological and psychiatric illness who are able to concentrate and to perform simple attention tasks are eligible.

Blind subjects: Early and late blind subjects (aged 18 to 80) will be included in this protocol.

Sighted subjects: Healthy sighted (normal or corrected-to normal vision) matched in age, sex, and handedness to the early blind subjects.

EXCLUSION CRITERIA:

Exclusion criteria for the study will be ny current medical or surgical condition or psychiatric or neurological illness.

Furthermore, any individual who is on medication with potential influence on nervous system function, who has a history of surgery with metallic implants or known history of metallic particles in the eye, cardiac pacemaker, intracardiac lines, neural stimulators, cochlear implants, pregnancy, or history of drug abuse will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45
Dates: Start 2004-01; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Amedi A, Malach R, Hendler T, Peled S, Zohary E. Visuo-haptic object-related activation in the ventral visual pathway. Nat Neurosci. 2001 Mar;4(3):324-30. doi: 10.1038/85201. PMID 11224551
- [Background] Amedi A, Raz N, Pianka P, Malach R, Zohary E. Early 'visual' cortex activation correlates with superior verbal memory performance in the blind. Nat Neurosci. 2003 Jul;6(7):758-66. doi: 10.1038/nn1072. PMID 12808458
- [Background] Bailes SM, Lambert RM. Cognitive aspects of haptic form recognition by blind and sighted subjects. Br J Psychol. 1986 Nov;77 ( Pt 4):451-8. doi: 10.1111/j.2044-8295.1986.tb02210.x. PMID 3801790